CLINICAL TRIAL: NCT01201902
Title: Randomized, Open, Clinical Study to Evaluate the Safety and Immunogenicity of an Inactivated Split-virion Influenza A(H1N1) Vaccine GC1116 With Adjuvant in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Immunogenicity of an Inactivated Split-virion Influenza A(H1N1) Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Medical Team, Green Cross Corparation
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GC1116; 임상제도과 - 649호(2009.9.28) (Registry Identifier: Korea Food & Drug Administraion)
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Influenza Infection
MeSH Terms: interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1 : Low dose with adjuvant (Experimental): Group 1: 18 ~ 64 years old subjects
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccine
- Group 1: High dose with adjuvant (Experimental): Group 1: 18 ~ 64 years old subjects
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccine
- Group1 : Plain vaccine (Active Comparator): Group 1: 18 ~ 64 years old subjects
  Interventions: Biological: un-adjuvanted influenza A(H1N1) vaccine
- Group 2 : Low dose with adjuvant (Experimental): Group 2: greater than or equal to 65 years of age
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccine
- Group 2 : high dose with adjuvant (Experimental): Group 2: greater than or equal to 65 years of age
  Interventions: Biological: Adjuvanted influenza A(H1N1) vaccine

INTERVENTIONS:
Biological: Adjuvanted influenza A(H1N1) vaccine — 0.25ml, Intramuscular on Day 0 and 21
  Other Names: Split-virion vaccine
  Arms: Group 1 : Low dose with adjuvant
Biological: Adjuvanted influenza A(H1N1) vaccine — 0.5ml, Intramuscular on Day 0 and 21
  Other Names: Split-virion vaccine
  Arms: Group 1: High dose with adjuvant
Biological: un-adjuvanted influenza A(H1N1) vaccine — 0.5ml, Intramuscular on Day 0 and 21
  Other Names: Split-virion vaccine
  Arms: Group1 : Plain vaccine
Biological: Adjuvanted influenza A(H1N1) vaccine — 0.25ml, Intramuscular on Day 0 and 21
  Other Names: Split-virion vaccine
  Arms: Group 2 : Low dose with adjuvant
Biological: Adjuvanted influenza A(H1N1) vaccine — 0.5ml, Intramuscular on Day 0 and 21
  Other Names: Split-virion vaccine
  Arms: Group 2 : high dose with adjuvant

SUMMARY:
The purpose of this study is to assess the safety and the body's immune response to an experimental H1N1 influenza vaccine in healthy adult and elderly populations. The study will enroll up to 590 healthy adults ages 18 and older with no history of H1N1 infection or vaccination. 354 individuals will be 18-64 years old, and the other 236 will be greater than or equal to 65 years of age.

DETAILED DESCRIPTION:
▶ Immunogenicity(Efficacy) Outcome Measures : Hemagglutination inhibition assay

1. Proportion of subjects, stratified by group, with seroconversion to HI antibody
2. Proportion of subjects, stratified by group, achieving a serum hemagglutination inhibition assay(HIA) antibody titer of 1:40 greater against the influenza H1N1 2009 virus
3. GMT(Geometric Mean Titer) and GMR(Geometric Mean Ratio) measuring by HIA antibody titer

   * Safety Outcome Measures :

1. Solicited adverse events(Day 0 ~ 6, Day 21 ~ 27) 2. Unsolicited adverse events(Day 0 ~ 42) 3. Adverse events(Day 21 ~ 6 months)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults age 18 and older.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Have a known allergy to eggs, chickens or other components of the vaccine(including MF59).
* Have immunosuppression including immunodeficiency disease.
* Have a history of Guillain-Barre Syndrome.
* Have a diagnosis of thrombocytopenia.
* Have a chronic disease that the investigator believes may interfere with successful completion of the study. (Excluding regulating hypertension)
* Hemophilia Patients or Are receiving anti-coagulating agents. Low-dose aspirin (100mg/day) purpose of prevention is allowed.
* Are receiving anti-viral agents.
* Have an acute fever, a temperature greater than 38℃(100.4 degrees Fahrenheit) within 72 hours of vaccination or Have a symptom of acute febrile illness within 14 days prior to vaccination in this study.
* Received below agents or expect to receive agents within following periods. A. Have immunosuppression therapy, radiotherapy, use of high-dose glucocorticoids or prednisolone(≥15mg/day) within 6 months prior to vaccination in this study.Inhaled, nasal and topical steroids are allowed) B. Have a history of receiving immunoglobulin or other blood product within 3 months prior to vaccination in this study.

C. Received an experimental agent within 1 month prior to vaccination in this study.

D. Received any vaccines(live licensed and inactivated licensed) within 1 month prior to vaccination in this study. (Excluding seasonal Influenza vaccine)

* Those who are not eligible to receive vaccine injection in the arm deltoid muscle.
* Pregnant females, Nursing mom, Those women who have a chance to become pregnant, but not taking a proper contraception.
* Not agree to abstain from drinking following 7 days of vaccination.
* Have any condition (clinically regardful medical or psychological condition) that would, in the opinion of the site investigator, render them unable to meet the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
HI antibody responses after 1 and/or 2 vaccinations | 21 days after vaccination

SECONDARY OUTCOMES:
Solicited local & general AE, Unsolicited AE, AE until 6 months after last vaccination | the date of vaccination until 6 days after vaccination, 42days after first vaccination, 6 months after last vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Woo-ju Kim, Principal Investigator — Korea University Guro Hospital